CLINICAL TRIAL: NCT04705909
Title: Efficacy of Statin Addition to Neoadjuvant Chemotherapy Protocols for Breast Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Omar Hamdy, Lecturer of Surgical oncology, Principal Investigator, Surgery department., Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2020 - 176
Record Dates: First submitted 2021-01-04; First posted 2021-01-12 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pitavastatin

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pitavastatin group (Experimental): For the intended neoadjuvant treatment period, participants will receive -in addition to standard chemotherapy protocol - Pitavastatin tablets 2 mg once daily.
  Interventions: Drug: Pitavastatin
- Placebo group (Placebo Comparator): For the intended neoadjuvant treatment period, participants will receive -in addition to standard chemotherapy protocol - Placebo tablets matching pitavastatin orally once daily.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Pitavastatin — Pitavastatin 2 mg oral tablets daily will be given to the patients concomitantly with the intended chemotherapy protocol for the treatment period prior to surgery.
  Other Names: HMG CoA reductase inhibitor " Lipovastatin"
  Arms: Pitavastatin group
Drug: placebo — patients in this group will receive placebo tablets concomitantly with the intended chemotherapy for the treatment period prior to surgery.
  Arms: Placebo group

SUMMARY:
Different modalities for breast cancer treatments have exhausting and distressing side effects and toxicities leading to decreased compliance. Thus, repurposing drugs with accepted safety profile and possible antitumor activity becomes an eminent constraint.

Statins have been reported to have possible advantages as anticancer, and control of cancer progression. Moreover, they can sensitize cancer cells for radiotherapy. Therefore, the investigators aim to investigate the effect of (pitavastatin) added to conventional chemotherapy protocols for breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent before any study-specific procedures.
* Histologic confirmation of invasive breast cancer.
* Plans for the administration of neoadjuvant chemotherapy.
* Not currently pregnant during the study

Exclusion Criteria:

* Severe gastrointestinal disorder
* Current use of statins or fibrates for any time during the 3 months before the study
* Proven hypersensitivity to statins
* Currently on medication for hypercholesterolemia
* Strong Cytochrome P450 3A4 (abbreviated CYP3A4) (e.g., clarithromycin, HIV protease inhibitors, and itraconazole), given potential interactions with statins
* Renal impairment with a creatinine > 1.4 mg/dl
* Hepatic impairment: Aspartate transaminase (AST)/(SGOT), Alanine Transaminase (ALT)/(SGPT) ≥ 2.5 x upper limit of the normal range (ULN), OR Total bilirubin ≥ 1.5 x ULN (subjects with Gilbert's syndrome can have bilirubin of up to 1.5 x ULN), OR Alkaline phosphatase > 2.5 x ULN
* Central nervous system (CNS) diseases and major psychiatric diseases or inability to comply with the protocol procedures
* Active infections
* Cardiac failure, class I-IV
* Current anticoagulant or antiplatelet aggregation therapy
* Current lactation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-01-15 (Estimated); Primary Completion 2021-09-15 (Estimated); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
clinical response rate | 6 months
  Response to preoperative therapy as per ultrasonographic tumor size assessment. A responder will have > 50% decrease in the size of the primary tumor without appearance of new lesions.
Relative reduction of Ki67 in tumor samples | 6 months
  It will be described as average pre-post differences in percent positive cells with 95% Wilson confidence intervals.

SECONDARY OUTCOMES:
The change in Cyclin D1 (candidate marker associated with breast tumor proliferation) | Baseline up to 6 months
The change in Cleaved caspase-3 (CC3) (candidate marker associated with tumor apoptosis) | Baseline up to 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of pharmacy, Mansoura university, Al Mansurah, Egypt

REFERENCES:
- [Derived] Dewidar SA, Hamdy O, Eltantawy A, El-Mesery M, El Gayar AM, Soliman MM. Effect of concomitant use of pitavastatin with neoadjuvant chemotherapy protocols in breast cancer patients: A randomized controlled clinical trial. Saudi Pharm J. 2022 Oct;30(10):1486-1496. doi: 10.1016/j.jsps.2022.07.011. Epub 2022 Jul 25. PMID 36387337